CLINICAL TRIAL: NCT00002282
Title: A Randomized Multicenter Study of the Efficacy, Safety, and Toleration of Fluconazole or Clotrimazole Troches in the Treatment of Patients With Oropharyngeal Candidiasis in Association With the Acquired Immunodeficiency Syndrome
Brief Title: A Comparison of the Safety and Effectiveness of Fluconazole or Clotrimazole in the Treatment of Fungal Infections of the Mouth and Throat in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012M; 056-171
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Fluconazole; Clotrimazole; Acquired Immunodeficiency Syndrome; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Clotrimazole; Fluconazole

INTERVENTIONS:
Drug: Clotrimazole
Drug: Fluconazole

SUMMARY:
To compare the efficacy, safety, and tolerance of fluconazole single daily capsule for 14 days versus clotrimazole troche 5 x daily for 14 days in the treatment of oropharyngeal candidiasis in patients with AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Cimetidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Known history of intolerance or allergy to imidazoles or triazoles, or the non-azole components of clotrimazole troches (dextrose, cellulose, povidone, magnesium stearate).
* Moderate or severe liver disease defined by specified lab values.

Concurrent Medication:

Excluded pending results of phase I studies to determine whether interaction between fluconazole and these agents occurs:

* Barbiturates.
* Phenytoin.
* Coumarin-type anticoagulants.
* Rifampin.
* Oral hypoglycemics.
* Cyclosporin.

Patients with the following are excluded:

* Known history of intolerance or allergy to imidazoles or triazoles, or the non-azole components of clotrimazole troches (dextrose, cellulose, povidone, magnesium stearate).
* Unable to tolerate oral medication.
* Moderate or severe liver disease defined by specified lab values.
* Life expectancy < 4 weeks.
* Unable or unwilling to be followed at the same center for the conduct of this study.

Prior Medication:

Excluded within 3 days of study entry:

* Other antifungal agents.
* Excluded pending results of phase I studies to determine whether interaction between fluconazole and these agents occurs:
* Barbiturates.
* Phenytoin.
* Coumarin-type anticoagulants.
* Rifampin.
* Oral hypoglycemics.
* Cyclosporin.

Patients meeting CDC criteria for diagnosis of AIDS, or having serologic or virologic evidence of HIV infection (but without AIDS-defining opportunistic infections as of yet).

* Patients who have given informed consent in writing to their participation in the study.
* Patients with signs of oropharyngeal candidiasis, i.e., with typical white plaques.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Dr Robert Larsen, Los Angeles, California
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - Davies Med Ctr, San Francisco, California
  - UCSF Hosp, San Francisco, California
  - Saint Raphael's Hosp, New Haven, Connecticut
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ Hosp, Boston, Massachusetts
  - Washington Univ School of Medicine, St Louis, Missouri
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Cabrini Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Ohio State Univ Hosp, Columbus, Ohio
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia